CLINICAL TRIAL: NCT06370052
Title: Pathophysiological Basis of Hidradenitis Suppurativa
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Sponsor
Other Study IDs: CHCRI-DJ-HS
Record Dates: First submitted 2024-03-20; First posted 2024-04-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- surgical procedure: HS patients, divided into three groups depending on the stage of hidradenitis, would participate in the study.
  The first and second groups would include stage 2-3 patients (according to the Hurley scale) in whom partial or complete clinical remission occurred after biological therapy and surgical treatment was performed according to the guidelines.
  In the third (control) group, we would classify the samples obtained from the above-mentioned patients, from whom we would take a sample of "normal" skin measuring 1 x 1 cm.
  GOAL: To determine the pathohistological changes in skin and subcutaneous tissues of patients with HS Hurley stage I and II and healthy patients (control group) and compare them with each other.
  Interventions: Procedure: excision

INTERVENTIONS:
Procedure: excision — excision of the affected area

SUMMARY:
HS is a chronic inflammatory disease manifested by recurrent inflammatory nodules, abscesses and tunnels under the skin. This disease is characterized by an inflammatory process that takes place in hair follicles, sebaceous glands and surrounding tissue. Because of its frequent recurrence and chronicity, it represents a major public health problem and there is a need for better diagnosis and new and more effective drugs. This research can be a part of realizing the stated needs.

DETAILED DESCRIPTION:
HS patients, divided into three groups depending on the stage of hidradenitis, would participate in the study.

The first and second groups would include stage 2-3 patients (according to the Hurley scale) in whom partial or complete clinical remission occurred after biological therapy and surgical treatment was performed according to the guidelines.

In the third (control) group, we would classify the samples obtained from the above-mentioned patients, from whom we would take a sample of "normal" skin measuring 1 x 1 cm.

With the standard procedure of pathohistological tissue processing after tissue fixation with 10% buffered formalin and embedding in paraffin, tissue sections stained with standard hematoxylin and eosin (HE) staining will be analyzed using a light microscope in such a way as to determine the type and amount of inflammatory infiltrate, the amount of granulation tissue and fibrosis and epithelial changes of the surface and follicular epithelium and graded according to intensity into 3 categories.

The mentioned tissue samples fixed in formalin and embedded in paraffin will be used to make tissue sections for immunohistochemical staining. The expression of inflammatory cytokines will be analyzed using the indirect peroxidase immunohistochemical method. Primary and secondary antibodies will be used for immunohistochemical analyses. The prepared tissue sections will be deparaffinized in a xylene solution and then dehydrated in a series of ethyl alcohols of decreasing concentrations (100%, 96% and 75%). It will then be washed three times with PBS solution and in citrate buffer (10mM, pH 6.0). Sections will then be washed with Triton X 100 solution (0.3% in PBS) at room temperature. After that, endogenous peroxidase will be inactivated using hydrogen peroxide in methanol (0.3%) for 30 minutes. After washing the tissue sections with PBS solution, normal serum (10%) will be added for 60 minutes. After washing the tissue sections in PBS solution (pH 7.4), the secondary antibody will be added depending on the primary one. Tissue rehydration will be done in ethyl alcohols of increasing concentrations (75%, 96% and 100%). After clarification with xylol, the preparation will be incorporated into entalan.

The intensity of immunohistochemical staining will be analyzed using the ImageJ computer program according to the staining intensity.

ELIGIBILITY:
Inclusion Criteria:

* Hidradenitis Suppurativa

Exclusion Criteria:

* patients with no HS
* patients who do not want to be in the clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiens with HS that are controlled in the region of CHC Rijeka
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The pathohistological changes | 24 months
  The pathohistological changes in skin and subcutaneous tissues of patients with HS Hurley stage I and II and healthy patients (control group) will be assessed and compared them with each other.

SECONDARY OUTCOMES:
The expression of cytokines | 24 months
  The expression of IL-1β, TNF-α, IL-8 and IL-10 by immunohistochemical method in skin and subcutaneous tissue of patients with HS Hurley stage II and III and healthy patients (control group) will be assessed and compared with each other
The correlation of the clinical Hurley classification and pathohistological changes | 12 months
  The clinical Hurley classification and pathohistological changes in the removed skin are meant to be correlated

CONTACTS AND LOCATIONS:
Overall Officials: Damir Juranić, MD, Principal Investigator — surgeon at CHC Rijeka

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: ICF
Time Frame: 24 months
Access Criteria: According to the GDPR, we will give the information to other researchers upon request under "label anonymous" just to preserve patients' identity.